CLINICAL TRIAL: NCT00276159
Title: Phase II Study of 852A Administered Subcutaneously in Patients With Hematologic Malignancies Not Responding to Standard Treatment
Brief Title: Study of Immune Response Modifier in the Treatment of Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug was not available.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05US02IMP-852A; MT2005-20 (Other: Blood and Marrow Transplantation Program); 2005LS057 (Other: Clinical Trials Office, University of Minnesota); 0509M73467 (Other: IRB, University of Minnesota); NCT00326937 (obsolete NCT alias)
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Results first posted 2010-05-05 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Multiple Myeloma; Chronic Lymphocytic Leukemia
Keywords: Leukemia; Lymphoma; Myeloma; Hematology; 852A; IRM; Oncology
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Neoplasms | interventions — N-(4-(4-amino-2-ethyl-1H-imidazo(4,5c)quinolin-1-yl)butyl)methanesulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 852A Treatment (Experimental): Patients receiving at least one dose of 852A.
  Interventions: Drug: 852A

INTERVENTIONS:
Drug: 852A — Subcutaneous injection 0.6 mg/m2 2 times/week/12 weeks, may increase by 0.2 mg/m2 up to 1.2 mg/m2.
  Other Names: Molecule 852A; S-32865

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity of 852A when used to treat certain hematologic malignancies not responding to standard treatment.

DETAILED DESCRIPTION:
852A will be administered as a subcutaneous injection (SC) 2 times per week for 12 weeks (24 doses) with provisions for dose escalation or reduction based on tolerability

ELIGIBILITY:
Subjects are eligible for the study if they meet all of the following

Inclusion Criteria:

* Diagnosis of one of the following hematologic malignancies not responding to at least 2 standard treatment regimens. Any criteria for persistent or recurrent disease acceptable, i.e. ≥5% blasts for acute leukemia.

  * acute lymphoblastic leukemia (ALL)
  * acute myeloid leukemia (AML)
  * non-Hodgkin's lymphoma (NHL)
  * Hodgkin's lymphoma (HL)
  * multiple myeloma (MM)
  * chronic lymphocytic leukemia (CLL)
* Performance status - Karnofsky > 50% for patients > 10 years of age or Lansky >50% for patients < 10 year of age
* Normal organ function within 14 days of study entry
* If female and of childbearing potential, are willing to use adequate contraception (hormonal, barrier method, abstinence) prior to study entry and for the duration of study participation. A female is considered to be of childbearing potential unless she has had her uterus removed, had a double oophorectomy, or has been amenorrheic for at least 6 months after chemotherapy

Exclusion Criteria:

* Had/have the following prior/concurrent therapy:

  * Systemic corticosteroids (oral or injectable) within 7 days of first dose of 852A (topical or inhaled steroids are allowed)
  * Investigational drugs/agents within 14 days of first dose of 852A
  * Immunosuppressive therapy, including cytotoxic agents within 14 days of first dose of 852A (nitrosoureas within 30 days of first dose)
  * Drugs known to induce QT interval prolongation and/or induce Torsades De Pointes unless best available drug required to treat life-threatening conditions
  * Radiotherapy within 4 weeks of the first dose of 852A
  * Hematopoietic cell transplantation 4 weeks of first dose of 852A
* Active infection or fever > 38.5°C within 3 days of first dose of 852A
* Cardiac ischemia, cardiac arrhythmias or congestive heart failure uncontrolled by medication
* History of, or clinical evidence of, a condition which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk
* Uncontrolled intercurrent or chronic illness
* Active autoimmune disease requiring immunosuppressive therapy within 30 days
* Active hepatitis B or C with evidence of ongoing viral replication
* Hyperthyroidism
* Uncontrolled seizure disorder
* Active coagulation disorder not controlled with medication
* Pregnant or lactating
* Concurrent malignancy (if in remission, at least 5 years disease free) except for localized (in-situ) disease, basal carcinomas and cutaneous squamous cell carcinomas adequately treated
* Proven active central nervous system (CNS) disease
* Human Immunodeficiency Virus (HIV) positive
* Congenital long QT syndrome or abnormal baseline QTc interval (> 450 msec in males and > 470 msec in females) after Bazett's correction (QTc msec = QT msec / square root of the RR interval in seconds) on screening electrocardiogram (ECG).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cooley, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 852A Treatment: Patients receiving at least 12 doses of 852A.
Period: Overall Study
Arm/Group | 852A Treatment
Started | 6
Completed | 0
Not Completed | 6
Not completed — Did not receive all 24 doses of 852A | 6

BASELINE CHARACTERISTICS:
Arm/Group | 852A Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (23.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 852A Response Using Modified Response Evaluation Criteria in Solid Tumors
Description: Stable disease in Non-Hogkin's Lymphoma = disease that does not satisfy complete (complete regression), partial (> or = 50% reduction) or progressive disease (increase of 25%) by at least a 4-week period. Since Acute Myelogenous Leukemia is not a solid tumor, Complete Response (CR) = <5% blasts with hematopoietic recovery (absolute neutrophil count >500) at 4 weeks.
Time Frame: Up to Week 12
Population: Includes patients receiving at least 12 doses of 852A study drug.
Measure: Number; unit: Participants
Arm/Group | 852A Treatment
Number analyzed (Participants) | 6
Participants
  Stable Disease | 1
  Partial Response | 1
  Progressive Disease | 4

2. Secondary Outcome: Number of Patients Who Received Steroids
Description: Number of patients who received steroids allowing successful continuation of therapy.
Time Frame: Up to Week 12
Population: Includes patients receiving at least 12 doses of 852A study drug.
Measure: Number; unit: Participants
Arm/Group | 852A Treatment
Number analyzed (Participants) | 6
Participants | 2

3. Secondary Outcome: Measure of Immune Activation With Correlative Laboratory Studies
Time Frame: Up to Week 12
Population: Analysis not done to sale of agent - unable to perform.
Arm/Group | 852A Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Peak Concentrations of 852A
Description: Measurement of peak concentrations of 852A to correlate the side effects of tolerability in patients.
Time Frame: Up to Week 12
Population: Not able to analysis due to sale of agent - unable to perform.
Arm/Group | 852A Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 of Treatment through Week 12
Arm/Group | 852A Treatment
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 852A Treatment (N=6)
Febrile neutropenia (Infections and infestations) | 1 (1)
Death (General disorders) | 2 (2) — Disease progression NOS
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 852A Treatment (N=6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema (Blood and lymphatic system disorders) | 1 (2)
Fatigue (General disorders) | 4 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Fever (General disorders) | 2 (4)
Chills (General disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (10)
Diaphoresis (Skin and subcutaneous tissue disorders) | 3 (3) — sweats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No